CLINICAL TRIAL: NCT04459897
Title: Lyon Granulomatous Hepatitis Study
Acronym: LGH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: LGH_2020
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Patient Diagnosed or Treated for Granulomatous Hepatitis Followed in the Internal Medicine (and or) Hepato-gastroenterology Departments
Keywords: Hepatitis Granulomatous; liver sarcoidosis; prognosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- diagnosed or treated for granulomatous hepatitis fol: The cohort is composed by patient diagnosed or treated for granulomatous hepatitis followed in the internal medicine and / or Hepato-gastroenterology departments (Croix-Rousse Hospital, Edouard-Herriot Hospital, Lyon Sud Hospital Center).
  Interventions: Other: Evaluation of epithelioid and gigantocellular granulomas within the hepatic parenchyma by histopathology approach.

INTERVENTIONS:
Other: Evaluation of epithelioid and gigantocellular granulomas within the hepatic parenchyma by histopathology approach. — : Retrospective histopathology review done by an expert of histopathology analysis (DAPI cell labeling). Analysis of the percentage of epithelioid cells and the percentage of gigantocellular granulomas in hepatic parenchyma of patient diagnosed for Hepatitis Granulomatous

SUMMARY:
Granulomatous hepatitis are histopathologically defined by the presence of epithelioid and gigantocellular granulomas within the hepatic parenchyma. Hepatic granulomas are observed in 2 to 15% of liver biopsies. Causes of granulomatous hepatitis can be related to ethnic and environmental factors and in western countries granulomatous hepatitis are mostly related to sarcoidosis and autoimmune cholangitis. Infections (mycobacteria, coxiella burnetii, hepatitis C) and medications also provide granulomatous hepatitis.

Sarcoidosis is a systemic disease of unknown etiology, which in third of cases has a chronic course. Five percent of patients die of their disease, mainly because of respiratory distress. Hepatic involvement is most often asymptomatic or pauci-symptomatic (moderate cholestasis and conglomerates of granulomas visible on imaging). More rarely, it can cause portal hypertension and its complications and be life-threatening.

The aim of the Lyon Hepatitis Granulomatous (LHG) study is to better characterize granulomatous hepatitis and within these, severe hepatic sarcoidosis. This is a retrospective study conducted from January 2008 to December 2016 proposed to all patients with granulomatous hepatitis followed in the internal medicine and / or Hepato-gastroenterology departments (Croix-Rousse Hospital, Edouard-Herriot Hospital, Lyon Sud Hospital Center). This study will cover 596 patients who had a liver biopsy showing granulomas.

The main objectives of the Lyon Hepatitis Granulomatous (LHG) study are to analyze i) the etiology of the disease and the contribution of molecular biology for infectious etiologies, ii) the contribution of nuclear imaging for sarcoidosis diagnosis versus conventional imaging, iii) treatment used and prognosis.

This study will permit a better characterization of granulomatous hepatitis, and liver sarcoidosis in terms of prognosis as well as therapeutic management.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of granulomatous hepatitis
* Patient followed in the internal medicine and / or Hepato-gastroenterology departments (Croix-Rousse Hospital, Edouard-Herriot Hospital, Lyon Sud Hospital Center)
* Collection of non-opposition

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient diagnosed or treated for granulomatous hepatitis followed in the internal medicine and / or Hepato-gastroenterology departments
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of epithelioid and gigantocellular granulomas within the hepatic parenchyma by histopathology approach. | at inclusion visit
  Retrospective histopathology review done by an expert of histopathology analysis (DAPI cell labeling). Analysis of the percentage of epithelioid cells and the percentage of gigantocellular granulomas in hepatic parenchyma of patient diagnosed for Hepatitis Granulomatous

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - : Hôpital de la Croix Rousse / GHN / service de médecine interne, Lyon
  - Hôpital Edouard Herriot / service de médecine interne, Lyon
  - Hôpital Lyon Sud / service de médecine interne, Pierre-Bénite